CLINICAL TRIAL: NCT00193895
Title: Post-operative Concurrent Chemo-radiotherapy Versus Post-operative Radiotherapy in High-risk Cutaneous Squamous Cell Carcinoma of the Head and Neck
Brief Title: Post-operative Concurrent Chemo-radiotherapy Versus Post-operative Radiotherapy for Cancer of the Head and Neck
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Princess Alexandra Hospital, Brisbane, Australia (Other); The Royal Australian and New Zealand College of Radiologists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 05.01
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Skin Cancer
Keywords: Skin cancer; radiotherapy; chemotherapy; surgery
MeSH Terms: conditions — Skin Neoplasms | interventions — Carboplatin; Injections; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiotherapy alone (Active Comparator): Radiotherapy alone (60Gy or 66Gy in 30-33 fractions 5-5/week)
  Interventions: Radiation: Radiotherapy
- Radiotherapy plus chemotherapy (Experimental): Radiotherapy plus chemotherapy (Radiotherapy 60Gy or 66Gy in 30-33 fractions 5/week + Carboplatin (AUC 2) intravenously weekly)
  Interventions: Drug: Carboplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will commence with a dose calculated to target an AUC of 2.0. A maximum of 6 doses of weekly Carboplatin will be given. Carboplatin will be administered intravenously over 20-30 minutes prior to radiation therapy.
  Other Names: Carboplatin Ebewe, Injection
  Arms: Radiotherapy plus chemotherapy
Radiation: Radiotherapy — 60 Gy OR 66Gy in 2Gy/fraction 5days/week
  Other Names: Radiation

SUMMARY:
The primary objective of the trial is to determine, in patients who have undergone surgery with curative intent for high-risk CSCC of the head and neck, whether there is a difference in time to loco-regional relapse between patients treated with post-operative concurrent chemo-radiotherapy ,consisting of Carboplatin, and post-operative radiotherapy alone. The target sample size for the trial is 266 patients and will take 3-4 years to accrue, based on an anticipated accrual of 80 patients/year. A further 2 years follow up is required.

DETAILED DESCRIPTION:
Two in every 3 Australians will be affected by skin cancer over their lifetime. The prevalence of skin cancer will continue to increase due to the ageing population and represents a significant problem in our community. Cure of early (T1-2) de novo cutaneous squamous cell carcinoma (CSCC) treated with either curative intent surgery or radiotherapy is 85-100%. However, the cure rate for locally advanced, recurrent, or metastatic disease to regional nodes following surgery alone are much lower, in the order of 20-70%. Metastatic CSCC is the most common malignancy of the parotid region in Australia. The 5 year loco-regional control with surgery alone is in the order of 40%-45%. The addition of post-operative radiotherapy improves loco-regional control by 15-20%, and is therefore considered the standard of care in this group of patients.

Recent data have shown that synchronous post-operative chemo-radiotherapy is superior to post-operative radiotherapy alone in "high-risk" mucosal head and neck squamous cell carcinoma (HNSCC). However, to date, there is no evidence from randomised trials that such a benefit exists in CSCC of the head and neck. At present there is little consensus amongst clinicians in Australia as to who should receive post-operative chemo-radiotherapy in CSCC. Although tumour control rates may be improved, the addition of chemotherapy may also significantly increase treatment related toxicity. Nonetheless, some centres have adopted the use of post-operative chemo-radiotherapy in selected patients with CSCC based on extrapolation from mucosal sites. This has resulted in a wide variability in practice for this disease.

Australia is uniquely placed to perform such a trial comparing post-operative chemo-radiotherapy to post-operative radiotherapy alone in high-risk CSCC due to the high rate of skin cancer. Currently there are limited data to guide management of patients with resected CSCC who are at high risk for recurrence. While it is reasonable to hypothesize that concurrent chemotherapy in this setting will confer a similar benefit to that seen in mucosal HNSCC, this can only be established by a randomized trial as proposed. If the addition of chemotherapy is shown to be beneficial and safe, then these results are likely to be translated into standard practice both nationally and internationally quite rapidly. On the other hand, if the treatment is found to be ineffective then patients will be spared the unnecessary toxicity and inconvenience associated with the addition of chemotherapy. A further important aspect of this trial will be the assessment of patient-related outcomes using a validated quality of life questionnaire. It will be important to ascertain whether any improvement in locoregional control due to the addition of chemotherapy, is also associated with improvement in quality of life compared to the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven SCC
* Patients have undergone either:

  * Resection of the primary lesion
  * Any type of parotidectomy (superficial, total, partial, etc.)
  * Any type of neck dissection(s)
* High risk feature(s); Advanced primary disease or high risk nodal disease

High Risk Nodal Disease

* Intra-parotid nodal disease (any number or size, with/without extracapsular extension, with/without an identifiable index lesion)
* Cervical nodal disease with a synchronous index lesion or previously resected cutaneous primary tumour (<5 years) within the corresponding nodal drainage and a mucosal primary has been excluded with at least a CT +/- MRI and panendoscopy* *For cervical nodal disease to be eligible there must be at least one of the following criteria:

  * > 2 nodes
  * largest node > 3 cm
  * Extracapsular extension

Advanced Primary Disease (TNM 6th Edition 2002) (Appendix 1)

* T3-4 primary disease (cartilage, skeletal, muscle, bone involvement, > 4 cm) of the head and neck including lip, nose and external auditory canal with or without nodal disease
* In transit metastases (metastases between the primary site and the adjoining nodal basin)

  * Age > 18 years
  * Written informed consent
  * ECOG <= 2
  * Absolute neutrophil count > 1.5 X 10^9/L, platelet count > 100 X 10^9/L, and haemoglobin > 10 g/dL (pre-radiotherapy blood transfusion to elevate the haemoglobin > 10 g/dL is permissible)
  * Calculated creatinine clearance (Cockcroft-Gault) >= 40 mL/min
  * Available for follow-up for up to 5 years
  * Life expectancy greater than 6 months

Exclusion Criteria:

* Intercurrent illness that will interfere with either the chemotherapy or radiotherapy such as immunosuppression due to medication or medical condition
* Metastasis(es) below the clavicles
* Previous radical radiotherapy to the head and neck, excluding treatment of an early glottic cancer greater than or equal to 2 years ago and superficial radiotherapy to cutaneous SCC or Basal cell carcinoma
* High risk for poor compliance with therapy or follow-up as assessed by investigator
* Pregnant or lactating women
* Patients with prior cancers, except: those diagnosed > 5 years ago with no evidence of disease recurrence and clinical expectation of recurrence of less than 5%; or successfully treated Level 1 cutaneous melanomas or early glottic cancer > 2 years ago; or non-melanoma skin cancer; or carcinoma in situ of the cervix.
* Low risk cervical nodal disease* without advanced primary disease

  *Low risk cervical nodal disease is defined as the presence of all of the following criteria:
* single nodal metastasis
* greater then or equal to 3cm,
* no extracapsular extension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2005-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Loco-regional Control | The date of primary outcome analysis will occur when the final patient has reached a minimum 2 years follow-up.

SECONDARY OUTCOMES:
Disease Free Survival | The date of analysis will occur when the final patient has reached a minimum 2 years follow-up.
Overall Survival | The date of analysis will occur when the final patient has reached a minimum 2 years follow-up.
Quality of Life | The date of analysis will occur when the final patient has reached a minimum 2 years follow-up.
Treatment-related Late Effects | The date of analysis will occur when the final patient has reached a minimum 2 years follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Porceddu, Study Chair — Princess Alexandra Hospital
Locations (21):
- Australia (17):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Riverina Cancer Centre, Wagga Wagga, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Illawarra Cancer Care Centre, Wollongong, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Brisbane Hospital, Herston, Queensland
  - Mater QRI, South Brisbane, Queensland
  - St Andrew's Toowoomba Hospital, Toowoomba, Queensland
  - North Queensland Oncology Service, Townsville, Queensland
  - Genesis Cancer Care (previously Premion), Tugun, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Andrew Love Cancer Care Centre, Geelong Hospital, Geelong, Victoria
  - William Buckland Radiotherapy Centre, The Alfred, Melbourne, Victoria
- New Zealand (4):
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Palmerston North Hospital, Palmerston North

REFERENCES:
- [Derived] Porceddu SV, Connolly E, Bressel M, Wratten C, Liu HY, Rischin D. Prognostic Subgroups for Disease-Free Survival With Cutaneous Squamous Cell Carcinoma of the Head and Neck: A Secondary Analysis of a Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2025 Oct 1;151(10):938-945. doi: 10.1001/jamaoto.2025.2110. PMID 40875250
- [Derived] Porceddu SV, Bressel M, Poulsen MG, Stoneley A, Veness MJ, Kenny LM, Wratten C, Corry J, Cooper S, Fogarty GB, Collins M, Collins MK, Macann AMJ, Milross CG, Penniment MG, Liu HY, King MT, Panizza BJ, Rischin D. Postoperative Concurrent Chemoradiotherapy Versus Postoperative Radiotherapy in High-Risk Cutaneous Squamous Cell Carcinoma of the Head and Neck: The Randomized Phase III TROG 05.01 Trial. J Clin Oncol. 2018 May 1;36(13):1275-1283. doi: 10.1200/JCO.2017.77.0941. Epub 2018 Mar 14. PMID 29537906
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au